CLINICAL TRIAL: NCT04237116
Title: A Randomized, Double-blind, Multicenter, 24-week Study of Subcutaneous Secukinumab to Assess Anti-interleukin-17A Treatment in Plaque Psoriasis Patients With Coexisting Non-alcoholic Fatty Liver Disease (pINPOINt)
Brief Title: A Study of Secukinumab Treatment in Patients With Plaque Psoriasis and Coexisting Non-alcoholic Fatty Liver Disease (NAFLD)
Acronym: pINPOINt
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457ADE15; 2019-003168-37 (EudraCT Number)
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Plaque Psoriasis; Non-alcoholic Fatty Liver Disease
Keywords: plaque psoriasis; NAFLD; NASH; PASI; secukinumab; non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: The primary objective of this study was to demonstrate superiority of secukinumab compared to placebo in patients with moderate to severe chronic plaque-type psoriasis and non-alcoholic fatty liver disease (NAFLD) with respect to psoriasis area and severity index (PASI) 90 response at Week 12.
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Arm - secukinumab (Experimental): secukinumab 300mg s.c. weekly in first 4 weeks, followed by q4w up to Week 20; and placebo 300mg s.c. at weeks 13, 14 and 15 to maintain the blind
  Interventions: Biological: Investigational Arm - secukinumab
- Control Arm - placebo (Placebo Comparator): placebo 300 mg s.c. weekly in first 4 weeks, followed by q4w up to Week 8; and secukinumab 300 mg s.c. weekly for 4 weeks starting at Week 12, followed by q4w up to Week 20
  Interventions: Biological: Control Arm - placebo

INTERVENTIONS:
Biological: Investigational Arm - secukinumab — secukinumab 300mg s.c. weekly in first 4 weeks, followed by q4w up to Week 20; and placebo 300mg s.c. at weeks 13, 14 and 15 to maintain the blind
  Other Names: AIN457
  Arms: Investigational Arm - secukinumab
Biological: Control Arm - placebo — placebo 300 mg s.c. weekly in first 4 weeks, followed by q4w up to Week 8; and secukinumab 300 mg s.c. weekly for 4 weeks starting at Week 12, followed by q4w up to Week 20
  Other Names: AIN457
  Arms: Control Arm - placebo

SUMMARY:
The aim of this study was to assess the therapeutic efficacy of secukinumab on the psoriatic skin and to explore the anti-inflammatory (reduction of hepatic inflammation and cell damage), anti-steatotic (reduction of hepatic triglyceride content) and anti-fibrotic (reduction of hepatic fibrosis) effects of secukinumab in patients with psoriasis and coexisting non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Primary outcome measure is Percentage of participants achieving ≥ 90% improvement (reduction) in PASI score compared to Baseline. Psoriasis Area and Severity Index (PASI) 90 response is defined as ≥ 90% improvement (reduction) in score compared to Baseline. It is a composite score where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. Score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. Primary analysis was planned to be performed comparing treatments with respect to the primary efficacy variable in a logistic regression model. It was planned to present the Odds Ratio and its 95%-confidence interval and p-value. Planned null hypothesis to be rejected was that the Odds Ratio of a PASI90 response for patients with secukinumab vs. patients with placebo is ≥1 after 12 weeks. Due to premature termination and limited number of treated patients with available data (7 in the secukinumab group and 3 in the placebo group), the extent of the originally planned statistical analyses of efficacy data was limited to descriptive summaries (absolute values per visit and changes from baseline; presented as mean and SD) for the score.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients, 18 years or older
* Moderate to severe plaque-type psoriasis, candidate for systemic therapy
* Diagnosis of NAFLD by either ultrasound at Screening or liver histology within 6 months before Baseline
* BMI > 25 kg/ m 2
* ALT 1.2 to 3.0 × ULN
* MRI confirmed Liver fat ≥ 8% at Screening

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type Psoriasis
* Drug induced psoriasis
* Pregnant or nursing (lactating) women
* Women of child bearing potential unless they are using effective methods of contraception
* Ongoing use of prohibited treatments
* Previous treatment with biological drug targeting IL-17 or the IL-17 receptor
* Past medical history record of infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C prior to Screening
* Unstable weight over the last 6 months prior to Screening.
* Type I diabetes, or uncontrolled diabetes (Type I or Type II) defined as HbAlc ≥ 10% at screening.
* Evidence of hepatic decompensation or severe liver impairment or cirrhosis
* History of liver transplantation or planned liver transplant or biliary diversion.
* Presence or history of other liver disease
* Current, or history of, significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening
* Prior or planned bariatric surgery
* Inability or unwillingness to undergo MRI of the abdomen
* Past medical history record of infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (7):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Plain Language Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 German centers and 1 Spanish center had randomized 8 and 2 patients, respectively.
  Patients who were still in the study when the sponsor terminated the study were counted as 'non-completers'.
Pre-assignment Details: This study was prematurely discontinued after the enrollment of 10 patients, because the recruitment was too slow to achieve the planned number of patients within a reasonable time frame. No safety issues led to the decision to terminate the study prematurely.
Period: Overall Study
Arm/Group | Investigational Arm - Secukinumab | Control Arm - Placebo
Started | 7 | 3
Completed | 3 | 1
Not Completed | 4 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Study terminated by Sponsor | 4 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Arm - Secukinumab | Control Arm - Placebo | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.8) | 32.0 (16.8) | 38.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 7 | 3 | 10

OUTCOME MEASURES:

1. Secondary Outcome: Serum Alanine Aminotransferase (ALT) Level
Description: ALT is an enzyme that the liver releases when it becomes inflamed or damaged. ALT level measures liver function Parameter.
  Normal range of values for ALT is about 7 to 56 units per liter (U/L). Higher levels of ALT in the blood indicate more liver problems.
  Due to the premature study termination and the limited number of treated patients with available data (7 patients in the secukinumab group and 3 patients in the placebo group), the extent of the originally planned statistical analyses of efficacy data was limited to descriptive summaries (absolute values per visit and changes from baseline; presented as mean and standard deviation) for the ALT score.
Time Frame: 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Investigational Arm - Secukinumab | Control Arm - Placebo
Number analyzed (Participants) | 7 | 3
U/L
  Baseline | 60.5 (35.73) | 89.0 (15.56)
  Week 12: number analyzed (Participants) | 4 | 2
  Week 12 | 43.3 (12.76) | 85.5 (20.51)

2. Secondary Outcome: Mean and SD of DLQI at Week 12
Description: Dermatology Life Quality Index (DLQI) is calculated by summing the score of each domain resulting in a maximum of 30 and a minimum of 0. The higher the score, the more Quality of Life was impaired. Meaning of DLQI Scores: 0-1 = no effect at all on patient's life, 2-5 = small effect on patient's life, 6-10 = moderate effect on patient's life, 11-20= very large effect on patient's life, 21-30 = extremely large effect on patient's life.
  Due to the premature study termination and the limited number of treated patients with available data (7 patients in the secukinumab group and 3 patients in the placebo group), the extent of the originally planned statistical analyses of efficacy data was limited to descriptive summaries (absolute values per visit and changes from baseline; presented as mean and standard deviation) for DLQI scores.
Time Frame: 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Investigational Arm - Secukinumab | Control Arm - Placebo
Number analyzed (Participants) | 7 | 3
Units on a scale
  Baseline | 11.3 (5.56) | 8.0 (8.49)
  Week 12: number analyzed (Participants) | 4 | 2
  Week 12 | 0.3 (0.50) | 7.0 (8.49)

3. Primary Outcome: Mean and SD Change From Baseline of PASI Score up to Week 12
Description: Psoriasis Area and Severity Index (PASI) 90 response is defined as ≥ 90% improvement (reduction) in score compared to Baseline. It is a composite score where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. Score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. Primary analysis was planned to be performed comparing treatments with respect to the primary efficacy variable in a logistic regression model.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS): Comprised all patients to whom study treatment/reference treatment had been assigned by randomization.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Investigational Arm - Secukinumab | Control Arm - Placebo
Number analyzed (Participants) | 7 | 3
Units on a scale
  Baseline (n=7,3) | 15.7 (4.22) | 15.9 (3.39)
  Week 12 (n=4,2): number analyzed (Participants) | 4 | 2
  Week 12 (n=4,2) | 0.8 (1.14) | 13.4 (0.35)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events were collected after signature of the informed consent form until 30 days after last dose of study treatment, and up to 24 weeks
Description: AEs and SAEs are any untoward sign or symptom that occurs during the study treatment and up to 24 weeks
Groups:
- Secukinumab 300mg: Secukinumab 300mg
- Placebo: Placebo
Arm/Group | Secukinumab 300mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/3
Other Adverse Events (participants affected / at risk) | 4/7 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300mg (N=7) | Placebo (N=3)
Aspartate aminotransferase increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300mg (N=7) | Placebo (N=3)
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Low density lipoprotein increased (Investigations) | 1 | 0
Urinary sediment abnormal (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to premature termination and limited number of treated patients (7 for secukinumab group and 3 in placebo), the extent of originally planned statistical analyses of efficacy was limited to descriptive summaries (absolute values per visit and changes from baseline; presented as mean and standard deviation) for the PASI score, ALT values, and DLQI scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT04237116/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04237116/SAP_001.pdf